CLINICAL TRIAL: NCT04248153
Title: An Exploratory Study to Determine the Optimal Timing of BR55 Contrast Enhanced Ultrasound (CEUS) of the Ovaries in Pre-menopausal Women
Brief Title: Optimal Timing of BR55 CEUS of the Ovaries
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision; expiration of available study agent due to long recruitment timeline.
Sponsor: Bracco Diagnostics, Inc (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BR55-109
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Group A: BR55 CEUS will be performed in the early follicular phase first and in the late follicular phase thereafter; Group B: BR55 CEUS will be performed in the late follicular phase first and in the early phase thereafter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): BR55 will be performed in the early follicular phase first and in the late follicular phase thereafter.
  Interventions: Drug: BR55
- Group B (Experimental): BR55 will be performed in the late follicular phase first and in the early follicular phase thereafter.
  Interventions: Drug: BR55

INTERVENTIONS:
Drug: BR55 — BR55 will be administered at doses of 0.03 mL/kg or 0.05 mL/kg

SUMMARY:
This is an exploratory, single center, open label, prospective study of BR55 to determine the optimal phase of the menstrual cycle for performing BR55 contrast-enhanced ultrasonography (CEUS) of the target ovary in premenopausal women scheduled to undergo preventative surgery because of high familial/hereditary or genetic risk for ovarian cancer.

ELIGIBILITY:
Inclusion Criteria: Enroll a subject in this study if the subject meets the following inclusion criteria:

* Is a female subject of at least 18 years of age;
* Is premenopausal;
* Is scheduled to undergo preventative salpingo-oophorectomy for high risk of ovarian cancer not earlier than 24 hours and not later than 5 days following the second BR55 CEUS examination;
* Provides written Informed Consent and is willing to comply with protocol requirements.

Exclusion Criteria: Exclude a subject from this study if the subject does not fulfill the inclusion criteria, or if any of the following conditions are observed:

* Is a pregnant or lactating female. Exclude the possibility of pregnancy:

  * by testing on site at the institution (serum βHCG) within 24 hours prior to the start of investigational product administration,
  * by surgical history (e.g., tubal ligation or hysterectomy),
* Has undergone prior systemic therapy for ovarian cancer;
* Has history of concurrent malignancy;
* Has history of any clinically unstable cardiac condition including class III/IV congestive heart failure;
* Has had any severe cardiac rhythm disorders within 7 days prior to enrolment;
* Has severe pulmonary hypertension (pulmonary artery pressure >90mmHg) or uncontrolled systemic hypertension and/or respiratory distress syndrome;
* Has open and/or non-healing wounds in the chest, abdomen and pelvis;
* Has other systemic vascular abnormalities associated with neovascularization that in the opinion of the investigator could significantly affect the ability to evaluate the effects of BR55;
* Is participating in a clinical trial or has participated in another trial with an investigational compound within the past 30 days prior to enrolment;
* Has previously been enrolled in and completed this study;
* Has any known allergy to one or more of the ingredients of the Investigational Product or to any other contrast media;
* Is determined by the Investigator that the subject is clinically unsuitable for the study;
* Has had major surgery, including laparoscopic surgery, within 3 months prior to enrolment;
* Has history of surgery to the ovaries or pelvic inflammatory disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subject of at least 18 years of age
Enrollment: 3 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luigia Storto, MD, Study Director — Bracco Diagnostics
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Up to 50 subjects were to be enrolled in the study: the first 3 as "training cases", the remaining divided between Group A and Group B.
Groups:
- Training Cases: Up to 3 subjects were to be enroll as "training cases" to determine the optimal imaging technique with BR55 and a 2D intracavitary probe for this study population. These subjects were to receive a single CEUS examination with administration of BR55 at a dose of 0.03 mL/kg, undergo all safety evaluations but not the efficacy assessments and were not required to undergo oophorectomy. Timing of the CEUS examination with respect to follicular phase of the menstrual cycle was not to be considered.
- Group A: BR55 will be performed in the early follicular phase first and in the late follicular phase thereafter.
  BR55: BR55 will be administered at doses of 0.03 mL/kg or 0.05 mL/kg
  No study participant was enrolled in this group.
- Group B: BR55 will be performed in the late follicular phase first and in the early follicular phase thereafter.
  BR55: BR55 will be administered at doses of 0.03 mL/kg or 0.05 mL/kg
  No study participant was enrolled in this group.
Period: Overall Study
Arm/Group | Training Cases | Group A | Group B
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The only participants enrolled in this study were 3 "training cases." No other study participant was enrolled in the study; therefore, there are no results for Group A and Group B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Training Cases | Group A | Group B | Total
Number analyzed (Participants) | 3 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 3 |  |  | 3
  >=65 years | 0 |  |  | 0
Age, Continuous [Mean (Full Range); unit: years] | 38.3 [35 to 43] |  |  | 38.3 [35 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  |  | 3
  Male | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 3 |  |  | 3
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  |  | 3
Actual Volume (mL) Injected [Mean (Full Range); unit: mL] | 2.06 [1.86 to 2.41] |  |  | 2.06 [1.86 to 2.41]

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of participants who received the contrast agent and experienced an adverse event.
Time Frame: From the time of signing Informed Consent through 24 hours post-dose, up to a maximum of 11 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Training Cases | Group A | Group B
Number analyzed (Participants) | 3 | 0 | 0
Participants | 0 |  |

ADVERSE EVENTS:
Time Frame: Safety monitoring was to begin at the time of signing Informed Consent through 24 hours post-dose, up to a maximum of 11 days.
Description: The only participants enrolled in this study were 3 "training cases." No other study participant was enrolled in the study; therefore, there are no results for Group A and Group B.
Arm/Group | Training Cases | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT04248153/Prot_SAP_000.pdf